CLINICAL TRIAL: NCT04515459
Title: Efficacy of Pre-operative Prehabilitation in Patients With Limb Sarcoma
Acronym: EPOP-SARCOMA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20 SARC 03
Record Dates: First submitted 2020-08-10; First posted 2020-08-17 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Sarcoma
Keywords: Bone sarcoma; Soft-tissue sarcoma; Pre-operative prehabilitation
MeSH Terms: conditions — Sarcoma; Bone Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients treated for bone or soft-tissue sarcoma of the limbs (Other)
  Interventions: Other: Surgical prehabilitation program.

INTERVENTIONS:
Other: Surgical prehabilitation program. — This programme will include the practice of general physical activity and the implementation of nutritional and psychological support.
  Each patient will have 8 Oncorehabilitation Transdisciplinary Evaluations (OTE):
  * 2 OTE will be performed before the surgery,
  * 6 OTE will be performed after the surgery.
  During the program (at each OTE), patients will also be asked to complete the QLQ-C30 questionnaire.

SUMMARY:
This Phase II feasibility study, prospective, interventional, monocentric aiming to assess the interest of pre-operative rehabilitation in patients treated for bone or soft-tissue sarcoma of the limbs.

This protocol will be based on the realisation of a surgical prehabilitation program adapted to the patient. This strategy will involve a team of several health professionals: rehabilitation doctor, physiotherapist, occupational therapist, specialised nurse, dietician and adapted physical activity teacher.

The aim of an adapted surgical prehabilitation program is to improve the functional recovery of the treated limb and the patient's autonomy after surgery.

Each patient will be followed until 24 months post surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age > or = 16 years old.
2. Patient with a diagnosis of bone or soft-tissue sarcoma confirmed by the "Réseau de Relecture en Pathologie Sarcomateuse (RRePS)"
3. Tumour localized in the lower or upper limb.
4. Localized or metastatic disease (in case of metastatic disease, the optimal surgical treatment for the primary tumor must be performed).
5. Indication of neoadjuvant treatment (radiotherapy and/or chemotherapy) according to the Multidisciplinary Concertation Meeting.
6. Inclusion before the initiation or during neoadjuvant treatment. In both cases, surgery must be scheduled between 6 and 10 weeks after inclusion, to permit the completion of the surgical prehabilitation.
7. Patient must provide written informed consent prior to any study-specific procedure. For minor patients, the holder(s) of parental authority must sign the informed consent and the patient's assent must be obtained.
8. Patient affiliated to the French social security system.

Exclusion Criteria:

1. Metastatic disease without optimal surgery planned of the primary tumour.
2. Any disease or medical condition that could interfere with study procedure, or that could, according to the judgment of investigator, expose the patient to an unacceptable risk.
3. Patient who has forfeited his/her freedom by administrative or legal award or who is under legal protection (curatorship and guardianship, protection of justice).
4. Any psychological, familial, geographic or social situation preventing compliance with the medical monitoring and/or with study procedure.
5. Pregnant or breastfeeding patient.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with a MSTS score (Musculoskeletal Tumor Rating Scale) greater than 75% at 24 months post-surgery. | 26 months for each patient.

SECONDARY OUTCOMES:
Quality of life using the Quality Of Life Questionnaire Core 30 (QLQ-C30). | 26 months for each patient.
  Quality of life will be evaluated from OTE1 to OTE8.
Anxiety using the Hospital Anxiety and Depression Scale (HADS). | 26 months for each patient.
  Seven item subscale. Each item is scored on a 4-point scale. Anxiety will be evaluated from OTE1 to OTE8.
Depression using the Hospital Anxiety and Depression Scale (HADS). | 26 months for each patient.
  Seven item subscale. Each item is scored on a 4-point scale. Depression will be evaluated from OTE1 to OTE8.
The patient functionality will be evaluated using the Tinetti's test from OTE1 to OTE8. | 26 months for each patient.
The patient functionality will be evaluated using the 6-min walk test from OTE1 to OTE8. | 26 months for each patient.
The patient functionality will be evaluated using the New Functional Ambulation Classification test from OTE1 to OTE8. | 26 months for each patient.
The patient functionality will be evaluated using the Box and Block Test from OTE1 to OTE8. | 26 months for each patient.
The patient functionality will be evaluated using the Frenchay Arm Test from OTE1 to OTE8. | 26 months for each patient.
The patient functionality will be evaluated using the Visual Analog Scale from OTE1 to OTE8. | 26 months for each patient.
The patient functionality will be evaluated using the Ricci and Gagnon's Score from OTE1 to OTE8. | 26 months for each patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse, France